CLINICAL TRIAL: NCT03794427
Title: Cognitive Changes After Hip Prosthesis; Comparison Between Combined Lumbosacral Nerve Block Versus Spinal Anesthesia: a Double Blind Randomized Clinical Trial
Brief Title: Combined Lumbosacral Nerve Block Versus Spinal Anesthesia for Cognitive Function After Hip Prothesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Anesthesiologist, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 181218
Record Dates: First submitted 2018-12-25; First posted 2019-01-07 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- unilateral lumbosacral nerve block (Experimental): Sciatic nerve block and paravertebral block at levels L3-L4 and L4-L5 will be performed
  Interventions: Other: unilateral lumbosacral nerve block; Other: Placebo at the spinal anesthesia level
- Spinal anesthesia (Active Comparator): spinal anesthesia will be performed
  Interventions: Other: Spinal anesthesia; Other: Placebo at lumbosacral level

INTERVENTIONS:
Other: unilateral lumbosacral nerve block — Patients will receive unilateral lumbosacral nerve block (sciatic nerve block and paravertebral block at levels L3-L4 and L4-L5). The sciatic nerve will be injected by 20 ml of the anesthetic mixture whereas levels L3-L4 and L4-L5 will be injected by a total of 20 ml of the anesthetic mixture without exceeding the maximum injected volume of 1 ml/kg.
  Arms: unilateral lumbosacral nerve block
Other: Spinal anesthesia — Patients will receive spinal anesthesia (3 ml of 0.5% bupivacaine)
  Arms: Spinal anesthesia
Other: Placebo at the spinal anesthesia level — Patients will receive 1 ml normal saline at the spinal anesthesia level (L3-L4 or L4-L5).
  Arms: unilateral lumbosacral nerve block
Other: Placebo at lumbosacral level — Patients will receive normal saline at the sciatic, L3-L4 and L4-L5 levels
  Arms: Spinal anesthesia

SUMMARY:
Hip fracture is a potentially devastating event, and serious surgical and medical complications occur frequently especially for elderly patients. Delirium is one of the common complications after hip surgery. Controversy exists regarding the possible impact of type of anesthesia (nerve block versus spinal) upon acute and long-term cognitive decline.

The primary objective is to assess the association between type of anesthesia (nerve block vs. spinal anesthesia) and risk of cognitive decline (CD). The secondary objective is to compare intra-operative hemodynamic changes, use of vasopressor drugs, and use of post-operative analgesics with respect to the type of anesthesia.

Prospective, double blind randomized clinical trial of hip fracture patients who will be assessed for CD pre- and postoperatively, using the Mini Mental State Examination (MMSE). The presence of CD will be determined at follow-up evaluation up to three months after surgery.

DETAILED DESCRIPTION:
Prospective, double blind randomized clinical trial of hip fracture patients who will be assessed for CD pre- and postoperatively, using the Mini Mental State Examination (MMSE). The presence of CD will be determined at follow-up evaluation up to three months after surgery. Patients undergoing hip surgery will be randomized into two groups. Group 1 will receive unilateral lumbosacral nerve block (sciatic nerve block and paravertebral block at levels L3-L4 and L4-L5) as well as placebo injection (1 ml normal saline) at the spinal anesthesia level (L3-L4 or L4-L5). The sciatic nerve will be injected by 20 ml of the anesthetic mixture whereas levels L3-L4 and L4-L5 will be injected by a total of 20 ml of the anesthetic mixture without exceeding the maximum injected volume of 1 ml/kg. Group 2 will receive spinal anesthesia (3 ml of 0.5% bupivacaine) in addition to placebo injection at the sciatic, L3-L4 and L4-L5 levels.

ELIGIBILITY:
Inclusion Criteria:

* Admitted with a hip fracture (femoral neck, trochanteric or sub-trochanteric)
* 40 kg in weight and higher

Exclusion Criteria:

Patients who are:

* Uncooperative
* Considered as moribund by the orthopedic surgeon at admission
* Alzheimer
* Severe cognitive impairment (MMSE<18)
* Absolute contraindication for spinal anesthesia (assessed preoperatively)
* Allergy to local anesthesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Cognitive decline | before operation (baseline)
  Patients' cognitive function will be assessed using the Mini Mental State Examination. The total score ranges between 0 and 30. A total score between 24 and 30 indicates no cognitive impairment. A score between 18 and 23 indicates mild cognitive impairment. A score between 0 and 17 indicates severe cognitive impairment
Cognitive decline | 1 day after the operation
  Patients' cognitive function will be assessed using the Mini Mental State Examination. The total score ranges between 0 and 30. A total score between 24 and 30 indicates no cognitive impairment. A score between 18 and 23 indicates mild cognitive impairment. A score between 0 and 17 indicates severe cognitive impairment
Cognitive decline | 7 days after the operation
  Patients' cognitive function will be assessed using the Mini Mental State Examination. The total score ranges between 0 and 30. A total score between 24 and 30 indicates no cognitive impairment. A score between 18 and 23 indicates mild cognitive impairment. A score between 0 and 17 indicates severe cognitive impairment
Cognitive decline | 1 month after the operation
  Patients' cognitive function will be assessed using the Mini Mental State Examination. The total score ranges between 0 and 30. A total score between 24 and 30 indicates no cognitive impairment. A score between 18 and 23 indicates mild cognitive impairment. A score between 0 and 17 indicates severe cognitive impairment
Cognitive decline | 2 months after the operation
  Patients' cognitive function will be assessed using the Mini Mental State Examination. The total score ranges between 0 and 30. A total score between 24 and 30 indicates no cognitive impairment. A score between 18 and 23 indicates mild cognitive impairment. A score between 0 and 17 indicates severe cognitive impairment
Cognitive decline | 3 months after operation
  Patients' cognitive function will be assessed using the Mini Mental State Examination. The total score ranges between 0 and 30. A total score between 24 and 30 indicates no cognitive impairment. A score between 18 and 23 indicates mild cognitive impairment. A score between 0 and 17 indicates severe cognitive impairment

SECONDARY OUTCOMES:
Intra-operative hemodynamic changes | 1 minute intra-operative
  Mean arterial pressure (in mmHg) will be recorded through a questionnaire
Intra-operative hemodynamic changes | 5 minutes intra-operative
  Mean arterial pressure (in mmHg) will be recorded through a questionnaire
Intra-operative hemodynamic changes | every 10 minutes intra-operative
  Mean arterial pressure (in mmHg) will be recorded through a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Naja, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon